CLINICAL TRIAL: NCT04943068
Title: A Phase 3, Bridging, Multicenter, Randomized, Double-blind, Placebo-controlled, Parallel-group Trial to Evaluate the Efficacy and Safety of Subcutaneously Administered Bremelanotide in Premenopausal Women With Hypoactive Sexual Desire Disorder (With or Without Decreased Arousal)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kwang Dong Pharmaceutical co., ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KD-BMT-301
Record Dates: First submitted 2021-06-10; First posted 2021-06-29 (Actual); Last update posted 2024-11-13 (Actual); Status verified 2024-11

CONDITIONS: Hypoactive Sexual Desire Disorder
Keywords: KD-BMT-301; Bremelanotide
MeSH Terms: conditions — Sexual Dysfunctions, Psychological | interventions — bremelanotide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Bremelanotide (Experimental): Bremelanotide (BMT) subcutaneously (SC) via auto-injector for 8-weeks double-Blind period
  Interventions: Drug: Bremelanotide
- Placebo (Placebo Comparator): Placebo subcutaneously (SC) via auto-injector for 4-weeks single-Blind period and for 8-weeks double-Blind period
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Bremelanotide — Subjects will self-administer a fixed dose (1.75 mg) of bremelanotide (BMT) subcutaneously (SC) via auto-injector.
  Arms: Bremelanotide
Drug: Placebo — Subjects will self-administer a Placebo subcutaneously (SC) via auto-injector.
  Arms: Placebo

SUMMARY:
The purpose of this study is to Evaluate the Efficacy and Safety of Subcutaneously Administered Bremelanotide in Premenopausal Women with Hypoactive Sexual Desire Disorder(with or without Decreased Arousal).

ELIGIBILITY:
[Main Inclusion Criteria]

* Has met diagnostic criteria for HSDD for at least 6 months
* Is willing and able to understand and comply with all study requirements
* Has a normal pelvic examination at screening

[Main Exclusion Criteria]

* Subjects should be generally healthy premenopausal females with no psychological, gynecological or urological conditions which might contribute to the sexual dysfunction, compromise study participation, or confound interpretation of the study results
* Not currently under treatment for the sexual dysfunction and willing to forego other treatments through the course of the clinical trial

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 193 (Actual)
Dates: Start 2021-05-10 (Actual); Primary Completion 2023-05-16 (Actual); Study Completion 2023-05-16 (Actual)

PRIMARY OUTCOMES:
Change from baseline to End of Study in the desire domain from the FSFI | Baseline up to End of Study(8weeks)

SECONDARY OUTCOMES:
Change from baseline to End of Study in FSDS-DAO (Item 13) | Baseline up to End of Study(8weeks)
Change from Baseline to End of Study in the Number of Satisfying Sexual Events (SSEs) Associated With Study Drug Administration | Baseline up to End of Study(8weeks)
Change from Baseline to End of Study in Mean Desire Score (Q3) From FSEP-R | Baseline up to End of Study(8weeks)
Change from Baseline to End of Study in Mean Satisfaction With Desire Score (Q4) From FSEP-R | Baseline up to End of Study(8weeks)
Change from Baseline to End of Study in the FSDS-DAO Total Score | Baseline up to End of Study(8weeks)
Change from Baseline to End of study in the total FSFI score based on the 19 questions | Baseline up to End of Study(8weeks)
  The FSFI total score is on a scale ranging from 2 to 36. Increasing scores on this scale represent an increase in sexual desire and is a positive outcome.
Change in mean Level of Sexual Arousal from FSEP-R Q6 | Baseline up to End of Study(8weeks)
Change in mean Satisfaction with Sexual Arousal from FSEP-R Q7. | Baseline up to End of Study(8weeks)
Change from Baseline to End of study in the scored time spent being concerned by difficulty with sexual arousal as measured by the FSDS-DAO Q14. | Baseline up to End of Study(8weeks)
Change from Baseline to End of study in the arousal domain from the FSFI Q3 through Q6. | Baseline up to End of Study(8weeks)
Change from Baseline to End of study in the total number of SSEs. | Baseline up to End of Study(8weeks)
Change from baseline in the desire domain from the FSFI Q1 and Q2 using all available double-blind data (visit 4, 5) | Baseline up to End of Study(8weeks)
Change from baseline in the score for feeling bothered by low sexual desire as measured by the FSDS -DAO Q13 using all available double-blind data(visit 4, 5) | Baseline up to End of Study(8weeks)
Change from baseline in the number of SSEs associated with study drug using the entire 8 weeks of the double-blind phase. | Baseline up to End of Study(8weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Soo Woong Kim, Dr, Principal Investigator — Seoul National University Hospital; Tak Kim, Dr, Principal Investigator — Korea University Anam Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea